CLINICAL TRIAL: NCT05324358
Title: A Randomized, Double-Blind, Double-Dummy, Parallel-Group, Active and Placebo-Controlled Trial to Evaluate the Analgesic Efficacy and Safety of NTM-001 for the Treatment of Moderately Severe Postoperative Pain Following Bunionectomy
Brief Title: Ketorolac Applied by Continuous IV Infusion for Treatment of Moderately Severe Postoperative Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neumentum, Inc. (Other)
Collaborators: NEMA Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NTM-001-CT001
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac Tromethamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NTM-001 Treatment Arm (Experimental): * NTM-001 loading dose of 12.5 mg administered over approximately 60 seconds, followed by a continuous IV infusion at a rate of 3.5 mg/h for 24h, by a pre-programmed infusion pump.
  * Subjects will also receive placebo to IV Morphine (injections).
  Interventions: Drug: Ketorolac Tromethamine; Other: IV Placebo for Morphine
- Morphine Treatment Arm (Active Comparator): * A single IV morphine bolus (4 mg) every 4h for up to 24h.
  * Subjects will also receive placebo to NTM-001.
  Interventions: Drug: Morphine Sulfate; Other: Intravenous Placebo for NTM-001
- Placebo Treatment Arm (Placebo Comparator): Subjects randomized will receive placebos of both active treatments concomitantly.
  * Placebo to NTM-001: Placebo "loading dose" applied over approximately 60 seconds, followed by a continuous IV infusion at a rate of 3.5 mL/h for 24h by a pre-programmed infusion pump.
  * Placebo to IV morphine injections: A single IV placebo bolus every 4h for up to 24h.
  Interventions: Other: Intravenous Placebo for NTM-001; Other: IV Placebo for Morphine

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Ketorolac tromethamine, alcohol free formulation, 1.0 mg/mL in saline solution (~0.9% NaCl) adjusted to a pH of ~7.4. Contained in a sterile, 200 mL polyolefin bag (filled with 125 mL of NTM-001).
  Other Names: NTM-001 (Ketorolac Tromethamine IV Continuous Infusion)
  Arms: NTM-001 Treatment Arm
Drug: Morphine Sulfate — Morphine single use vials at 4 mg/mL, filled with 1 mL.
  Other Names: Morphine Sulfate Injection USP
  Arms: Morphine Treatment Arm
Other: Intravenous Placebo for NTM-001 — Placebo alcohol free saline solution (~0.9% NaCl; matching active NTM-001). Contained in a sterile, 200 mL polyolefin bag (filled with 125 mL Placebo solution).
  Arms: Morphine Treatment Arm; Placebo Treatment Arm
Other: IV Placebo for Morphine — Placebo single use vials with saline (matching active morphine).
  Arms: NTM-001 Treatment Arm; Placebo Treatment Arm

SUMMARY:
This clinical study is a randomized, double-blind, double-dummy, parallel group, multi-center, active and placebo-controlled trial evaluating the analgesic efficacy and safety of NTM-001 in subjects with moderately severe postoperative pain after bunionectomy surgery.

This study is designed to compare the efficacy of NTM-001 to placebo. Intravenous (IV) morphine serves as an active comparator to determine assay sensitivity and support assessment of opioid-level analgesia for NTM-001. Effectiveness, safety, and tolerability parameters will be descriptively compared between treatment arms.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed.
2. Male or female subjects between 18 and <65 years of age at time of consent.
3. Body weight ≥50 kg.
4. Physical status rated as ≤2 on the American Society of Anesthesiologists (ASA) rating scale (Owens, Felts et al. 1978).
5. Scheduled to undergo primary unilateral first metatarsal bunionectomy.
6. Women must be postmenopausal, surgically sterile, abstinent, or practicing or agree to practice an effective method of birth control if they are sexually active before entry, throughout the study, and for 7 days after the last dose of study drug (effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier method, and male partner sterilization). Women of childbearing potential must have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test at screening and a negative urine pregnancy test before surgery.
7. Subject is willing and able to complete all study procedures including training on pain scales, follow instructions, communicate meaningfully with study personnel, and return for all visits as listed in the protocol.

Exclusion Criteria:

1. History of peptic ulcer disease, GI bleeding, perforation, or active peptic ulcer disease.
2. History of asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs.
3. History of, or suspected or confirmed, cerebrovascular bleeding, hemorrhagic diathesis, or incomplete hemostasis.
4. Increased risk of bleeding at the discretion of the Investigator based on prior/concomitant disease, laboratory values, medication or surgical complications.
5. Clinical laboratory values reflecting at least mild renal insufficiency as indicated by a creatinine clearance ≤89 mL/min.
6. Risk for renal failure due to volume depletion at the discretion of the Investigator.
7. Concomitant use of aspirin or NSAIDs.
8. History of seizure disorder or epilepsy, as suggested by the presence of any of the following:

   * Mild or moderate traumatic brain injury, stroke, transient ischemic attach, or brain neoplasm within 1 year of screening.
   * Severe traumatic brain injury, episode(s) of unconsciousness of more than 24 hours duration, or posttraumatic amnesia of more than 24 hours duration within 15 years of screening.
9. History of alcohol or drug abuse in the Investigator's judgement based on subject history and physical examination.
10. Significant chronic obstructive pulmonary disease or cor pulmonale, a substantially decreased respiratory reserve, hypoxia, hypercapnia, or pre-existing respiratory depression.
11. At least moderately impaired hepatic function (Child-Pugh >6), or subjects with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values greater than 3 times the upper limit of normal (ULN).
12. Concurrent use of monoamine oxidase inhibitors (MAOIs) or use of MAOIs within the last 14 days.
13. The subject is not on a stable dose (at least 2 weeks prior to Screening Visit) of medications that may lower the seizure threshold (e.g., anti-psychotic agents) or which impact the serotonergic system (e.g., selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants).
14. Evidence of significant anemia (indicated by hemoglobin concentration ≤8 g/dL).
15. Evidence of active infections that may spread to other areas of the body (e.g., osteomyelitis, pyogenic infection of the hip, Hepatitis B or C, or other overt infections) or a history of human immunodeficiency virus (HIV) 1 or 2.
16. History of malignancy within 2 years prior to the start of the study, with the exception of basal cell and cutaneous squamous cell carcinoma.
17. History of systemic lupus erythematosus, antiphospholipid syndrome, vasculitis, vasculopathy, or deep vein thrombosis.
18. Uncontrolled or poorly controlled post-traumatic stress disorder, generalized anxiety disorder, depression, psychiatric, or other significant medical conditions.
19. Chronic systemic steroid therapy, excluding inhalers or a 1-time intraoperative dose, within 4 weeks before screening.
20. History of pending litigation due to pain or disability.
21. Clinically significant disease that, in the Investigator's opinion, may affect efficacy or safety assessments.
22. Employees of the Investigator or study site with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, including family members of the employees or the Investigator.
23. Received an experimental drug or used an experimental medical device within 30 days before screening or have participated in a previous study of ketorolac.
24. Contraindications to, or history of allergy or hypersensitivity to ketorolac and/or morphine and their excipients.
25. A positive COVID-19 test (rapid antigen test) or COVID-19 related symptoms at screening and/or at check in of Visit 2 (Surgical Period).
26. Subjects who are planning on receiving a COVID-19 vaccine during the study duration.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 341 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference (SPID24) | 0 to 24 hours after start of administration
  The primary endpoint is the Summed Pain Intensity Difference over 24h (SPID24) from start to end of administration of investigational medicinal product (IMP). Calculated as the weighted sum of the PID (difference between baseline at qualifying period and current pain intensity) collected at protocol scheduled time points through up to 24h after starting infusion of the IMP, using the following formula: SPID24 = Σ Wi * PIDi (1) where the Σ sums over all observations collected from the first assessment after the first IMP administration to Hour 24 and Wi is the time elapsed from the previous observation PIDi-1 to the current observation PIDi.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Sun City Clinical Research, Sun City, Arizona
  - Trovare Clinical Research, Bakersfield, California
  - Alliance Research Intitute, Canoga Park, California
  - Pasadena Clinical Trials, Pomona, California
  - Dr. Vince Clinical Research, Overland Park, Kansas
  - Chesapeake Research, Pasadena, Maryland
  - Curalta Clinical Trials, Westwood, New Jersey
  - Midwest Clinical Research Center, Dayton, Ohio
  - The Orthopedic Center, Tulsa, Oklahoma
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No